CLINICAL TRIAL: NCT03490383
Title: ERCP Based Study of Microbiota in Bile From Patients With Common Bile Duct Stone
Brief Title: Study of Microbiota in Bile From Patients With Common Bile Duct Stone During ERCP
Status: Completed | Type: Observational
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhaohang, Dr., Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: CBD stone and microbiota
Record Dates: First submitted 2018-03-14; First posted 2018-04-06 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Common Bile Duct Calculi; Microbial Colonization
Keywords: ERCP; CBD stone; Microbial Colonization
MeSH Terms: conditions — Gallstones; Communicable Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients without CBD calculi: patients without CBD calculi
- CBD calculi without ERCP history: patients with CBD calculi without ERCP history
- CBD calculi with ERCP history: patients with CBD calculi and ERCP history

SUMMARY:
In this study, investigators will investigate the microbiota of bile in common bile duct stone participants. Three key questions are of concern. The first one is whether there is bacteriria in bile in participants without common bile duct stone. The second one is whether the microbiota of bile is similar with that of gut mucosa in common bile duct stone participants. The third one is whether the bacteria in bile of common bile participants with intact papillar is the same as that of participants underwent sphinctomy.

ELIGIBILITY:
Inclusion Criteria:

* CBD tumor or CBD calculi

Exclusion Criteria:

* contraindication for ERCP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ERCP patients in our center
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
microbiota in bile | intraoperative
  16s RNA

CONTACTS AND LOCATIONS:
Overall Officials: Hang Zhao, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Shang General Hospital, Shanghai
  - Shanghai Municipal Hospital of Traditional Chinese Medicine, Shanghai